CLINICAL TRIAL: NCT03847428
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Multi Center Study of Durvalumab Monotherapy or in Combination With Bevacizumab as Adjuvant Therapy in Patients With Hepatocellular Carcinoma Who Are at High Risk of Recurrence After Curative Hepatic Resection or Ablation
Brief Title: Assess Efficacy and Safety of Durvalumab Alone or Combined With Bevacizumab in High Risk of Recurrence HCC Patients After Curative Treatment
Acronym: EMERALD-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D910DC00001; 2023-507689-26-00 (Registry Identifier: CTIS); 2018-004105-85 (EudraCT Number)
Record Dates: First submitted 2019-02-18; First posted 2019-02-20 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Early stage HCC; Durvalumab; Bevacizumab; Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — durvalumab; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Durvalumab 1120 mg (Q3W) + bevacizumab 15 mg/kg (Q3W)
  Interventions: Drug: Durvalumab; Drug: Bevacizumab
- Arm B (Experimental): Durvalumab 1120 mg (Q3W) + bevacizumab placebo (Q3W)
  Interventions: Drug: Durvalumab; Other: Placebo
- Arm C (Placebo Comparator): Durvalumab placebo (Q3W) + bevacizumab placebo (Q3W)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Durvalumab — Durvalumab IV (intravenous)
  Other Names: IMFINZI
  Arms: Arm A; Arm B
Drug: Bevacizumab — Bevacizumab IV (intravenous)
  Other Names: AVASTIN
  Arms: Arm A
Other: Placebo — Saline solution for Durvalumab and/or Bevacizumab masking (IV intravenous) or Dextrose for Durvalumab masking
  Arms: Arm B; Arm C

SUMMARY:
A global study to assess the efficacy and safety of durvalumab in combination with bevacizumab or durvalumab alone in patients with hepatocellular carcinoma who are at high risk of recurrence.

DETAILED DESCRIPTION:
This is a Phase III, randomized, double-blind, placebo-controlled, multi-center, global study to assess the efficacy and safety of durvalumab in combination with bevacizumab or durvalumab monotherapy or placebo as adjuvant therapy. This study will be conducted in patients with HCC who are at high risk of recurrence after curative hepatic resection or ablation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically (or radiologically for patients undergoing curative ablation), newly diagnosed, confirmed HCC and successfully completed curative therapy (resection or ablation)
* Imaging to confirm disease-free status within 28 days prior to randomization
* ECOG 0-1 at enrolment
* Child-Pugh score of 5 or 6
* Adequate organ and marrow function.

Exclusion Criteria:

* Known fibrolamellar HCC, sarcomatoid HCC or mixed cholangiocarcinoma and HCC
* Evidence of metastasis, macrovascular invasion or co-existing malignant disease on baseline imaging
* History of hepatic encephalopathy within 12 months prior to randomization
* Evidence, by Investigator assessment, of varices at risk of bleeding on upper endoscopy or contrast-enhanced cross-sectional imaging
* Patients with Vp1 to Vp4 portal vein thrombosis on baseline imaging are excluded
* Active co-infection with HBV and HDV.
* Receipt of prior systemic anticancer therapy for HCC
* Those on a waiting list for liver transplantation

Ages: 18 Years to 150 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 908 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2026-05-29 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival (RFS) for Arm A vs Arm C | Up to 49 months after first patient randomized
  RFS (per RECIST 1.1 criteria as assessed by BICR) will be defined as the time from the date of randomization until the date of the first objective radiologic recurrence or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Recurrence-free survival (RFS) Arm B vs Arm C | Up to 49 months after first patient randomized
  RFS (per RECIST 1.1 criteria as assessed by BICR) will be defined as the time from the date of randomization until the date of the first objective radiologic recurrence or death due to any cause, whichever occurs first.
Overall Survival (OS) for Arm A vs Arm C and Arm B vs Arm C | No timeframe
  OS is defined as the time from the date of randomization until death due to any cause
Recurrence-free survival at 24 months (RFS24) and 36 months (RFS36) for Arm A vs Arm C and Arm B vs Arm C | At 24 and at 36 months
  Proportion of RFS at 24 months and at 36 months
Time to recurrence (TTR) for Arm A vs Arm C and Arm B vs Arm C | Up to 49 months after first patient randomized
  TTR is defined as the time from the date of randomization until the date of disease recurrence
Time from randomization to recurrence/progression on next therapy (RFS2/PFS2) for Arm A vs Arm C and Arm B vs Arm C | Up to 49 months after first patient randomized
  Time from randomization to recurrence/progression on next therapy (RFS2/PFS2)

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, PhD, Principal Investigator — Liver Cancer Institute Zhongshan Hospital, Fudan University; Jennifer Knox, MD, Principal Investigator — Solid Tumor Medical Oncology Princess Margaret Cancer Centre
Locations (173):
- United States (34):
  - Research Site, Birmingham, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Costa Mesa, California
  - Research Site, La Jolla, California
  - Research Site, Long Beach, California
  - Research Site, Orange, California
  - Research Site, Sacramento, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Miami, Florida
  - Research Site, Tampa, Florida
  - Research Site, Honolulu, Hawaii
  - Research Site, Chicago, Illinois
  - Research Site, Westwood, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Shreveport, Louisiana
  - Research Site, Detroit, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Omaha, Nebraska
  - Research Site, New Brunswick, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, New York, New York
  - Research Site, Stony Brook, New York
  - Research Site, Durham, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Spartanburg, South Carolina
  - Research Site, Knoxville, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Madison, Wisconsin
- Australia (4):
  - Research Site, Kogarah
  - Research Site, Melbourne
  - Research Site, Nedlands
  - Research Site, Westmead
- Austria (3):
  - Research Site, Innsbruck
  - Research Site, Linz
  - Research Site, Sankt Pölten
- Brazil (7):
  - Research Site, Florianópolis
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Santa Maria
  - Research Site, Santo André
  - Research Site, São José do Rio Preto
  - Research Site, Vitória
- Canada (5):
  - Research Site, Hamilton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Québec, Quebec
- China (19):
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Hohhot
  - Research Site, Nanjing
  - Research Site, Ningbo
  - Research Site, Shanghai
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Zhengzhou
- Egypt (6):
  - Research Site, Alexandria
  - Research Site, Asyut
  - Research Site, Cairo
  - Research Site, Dakahlia
  - Research Site, New Cairo
  - Research Site, Shebeen El Kom
- France (11):
  - Research Site, Amiens
  - Research Site, Angers
  - Research Site, Besançon
  - Research Site, Clichy
  - Research Site, Dijon
  - Research Site, Nantes
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Toulouse
  - Research Site, Tours
- Germany (10):
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Chemnitz
  - Research Site, Cologne
  - Research Site, Freiburg im Breisgau
  - Research Site, Heidelberg
  - Research Site, Leipzig
  - Research Site, Lübeck
  - Research Site, München
  - Research Site, Tübingen
- Hong Kong (3):
  - Research Site, Hong Kong
  - Research Site, Kwai Chung
  - Research Site, Shatin
- India (5):
  - Research Site, Bangalore
  - Research Site, Hyderabad
  - Research Site, Kolkata
  - Research Site, Mumbai
  - Research Site, New Delhi
- Italy (6):
  - Research Site, Bologna
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Roma
  - Research Site, Tricase, Lecce
  - Research Site, Verona
- Japan (24):
  - Research Site, Bunkyō City
  - Research Site, Fukuoka
  - Research Site, Gifu
  - Research Site, Hiroshima
  - Research Site, Kōtoku
  - Research Site, Kumamoto
  - Research Site, Kurume-shi
  - Research Site, Kyoto
  - Research Site, Matsuyama
  - Research Site, Mitaka-shi
  - Research Site, Musashino-shi
  - Research Site, Nagasaki
  - Research Site, Nagoya
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shinagawa-ku
  - Research Site, Shinjuku-ku
  - Research Site, Shiwa-gun
  - Research Site, Takasaki-shi
  - Research Site, Tsu
  - Research Site, Wakayama
  - Research Site, Yokohama
- Peru (2):
  - Research Site, Lima
  - Research Site, San Isidro
- Philippines (3):
  - Research Site, City of Muntinlupa
  - Research Site, Manila
  - Research Site, Pasig
- Poland (4):
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Poznan
  - Research Site, Warsaw
- Research Site, Ponce, Puerto Rico
- Russia (5):
  - Research Site, Barnaul
  - Research Site, Moscow
  - Research Site, Obninsk
  - Research Site, Saint Petersburg
  - Research Site, Yekaterinburg
- Research Site, Singapore, Singapore
- South Korea (3):
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Seoul
- Taiwan (5):
  - Research Site, Changhua
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan
  - Research Site, Yunlin
- Thailand (5):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Pathum Thani
- Turkey (Türkiye) (4):
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Malatya
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home